CLINICAL TRIAL: NCT06661070
Title: Short-term Effectiveness of High- and Low-intensity Percutaneous Electrolysis in Patients With Low Back Pain
Brief Title: Electrolysis in Patients With Low Back Pain
Acronym: Electrolysis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Collaborators: Universidad Complutense de Madrid (Other); Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Sebastian Klich, Principal Investigator, Wroclaw University of Health and Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCM#1; #19/044 (Other: Clinical Ethics Committee of Hospital Clínico San Carlos)
Record Dates: First submitted 2024-10-18; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Low Back Pain
Keywords: Low Back; Pain; Multifidus muscle; Trigger Points; shear-wave elastography; pain sensitivity
MeSH Terms: conditions — Low Back Pain; Pain | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: A triple-blinded, pilot randomized controlled trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-intensity percutaneous electrolysis (HIPE) (Experimental): The HIPE group receives a 660 mA galvanic current for 10 s.
  Interventions: Device: Electrolysis Percutaneous Therapeutic (EPTE)
- Low-intensity percutaneous electrolysis (LIPE) (Experimental): The LIPE group receives a 220 mA × 30 s.
  Interventions: Device: Electrolysis Percutaneous Therapeutic (EPTE)
- Dry Needling (DN) (Active Comparator): The DN group received no galvanic current.
  Interventions: Other: Dry Needling

INTERVENTIONS:
Device: Electrolysis Percutaneous Therapeutic (EPTE) — EPTE device (Ionclinics, Valencia, Spain)
  Arms: High-intensity percutaneous electrolysis (HIPE); Low-intensity percutaneous electrolysis (LIPE)
Other: Dry Needling — A dry needle with size 0.30 × 40 (Agupunt, Barcelona, Spain)
  Arms: Dry Needling (DN)

SUMMARY:
The goal of this observational study is to investigate the efficacy of percutaneous electrolysis compared with dry needling on pain sensations and multifidus muscle properties in subjects with low back pain. The main questions it aims to answer are:

The high-intensity and low-intensity percutaneous electrolysis may induce pressure pain threshold (PPT) changes in myofascial trigger points in the low back during the intervention compared with dry needling.

Percutaneous electrolysis interventions may reduce stiffness in the multifidus muscle during the intervention compared with dry needling.

DETAILED DESCRIPTION:
A parallel-group, controlled, triple-blinded, randomized pilot clinical trial comparing the effects of a single session of high-intensity percutaneous electrolysis (HIPE), low-intensity percutaneous electrolysis (LIPE), and dry needling (DN) applied to the multifidus muscle most active MTrP in subjects with low back pain. This clinical trial will follow the Consolidated Standards of Reporting Trials for pragmatic clinical trials.

This procedure consists of three trials, i.e., (1, HIPE) 660 uA x 30"; (2, LIPE) 220uA x 30"; and (3, DN) with 1 twitch response, and the needle inserted 30".

ELIGIBILITY:
Inclusion Criteria:

* to report low back pain of at least six months duration,
* aged 35 to 50 years,
* at least one active trigger point is present in the multifidus muscle.

Exclusion Criteria:

* pharmacological (e.g., analgesics) or physiotherapy treatment before or during their participation in the study,
* needle fear,
* prior lower extremity or spine surgery, absence of pain, any musculoskeletal or neuropathic conditions (e.g., peripheral compressive neuropathy, radiculopathy, sarcopenia, fibromyalgia, muscle ruptures), traumatic injuries (e.g., fractures or fissures), or any medical condition or contraindication for needling treatment (e.g., anticoagulants).

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-04 (Estimated); Primary Completion 2024-11-23 (Estimated); Study Completion 2024-11-23 (Estimated)

PRIMARY OUTCOMES:
Pain changes in pain intensity before and after the intervention | Baseline, immediately after, and 24 after of intervention
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) will be used to assess the patient's current level of shoulder pain, and the worst and lowest level of pain experienced in the preceding week in the shoulder area.

SECONDARY OUTCOMES:
Pressure Pain Threshold | Baseline, immediately after, and 24 after of intervention
  Somedic Algometer type 2 was used to measure PPT. The diameter of the contact tip was 10 mm and covered with 2 mm thick rubber. The pressure on point and its rate was standardized (30 kPa s-1 ). The value of the pain threshold equals the value of the pressure at which the examined person reported that the pressure exerted on a certain point causes pain.
Muscle stiffness | Baseline, immediately after, and 24 after of intervention
  An ultrasound machine with shear-wave elastography Canon Aplio A device, using a linear transducer PLT-1005-BT (Canon Medical Corp, 1385 Shimoishigami, Otawara, Tochigi 324-8550, Japan). The console settings will also be standard for all the acquisitions (Frequency=11 MHz, Gain=78 dB, Dynamic Range=75, and Depth=4.5 cm).

CONTACTS AND LOCATIONS:
Overall Officials: Juan Antonio Valera-Calero, PhD, Study Director — Universidad Complutense de Madrid
Locations (1):
- Faculty of Nursery, Physiotherapy and Podiatry, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rozenfeld E, Finestone AS, Moran U, Damri E, Kalichman L. Test-retest reliability of myofascial trigger point detection in hip and thigh areas. J Bodyw Mov Ther. 2017 Oct;21(4):914-919. doi: 10.1016/j.jbmt.2017.03.023. Epub 2017 Mar 29. PMID 29037648
- [Result] Fernandez-de-Las-Penas C, Dommerholt J. International Consensus on Diagnostic Criteria and Clinical Considerations of Myofascial Trigger Points: A Delphi Study. Pain Med. 2018 Jan 1;19(1):142-150. doi: 10.1093/pm/pnx207. PMID 29025044
- [Result] Valera-Calero JA, Sanchez-Mayoral-Martin A, Varol U. Short-term effectiveness of high- and low-intensity percutaneous electrolysis in patients with patellofemoral pain syndrome: A pilot study. World J Orthop. 2021 Oct 18;12(10):781-790. doi: 10.5312/wjo.v12.i10.781. eCollection 2021 Oct 18. PMID 34754834